CLINICAL TRIAL: NCT04293250
Title: Preoperative Moderate-to-vigorous Intensity Physical Activities Reduce Postoperative Pain in Adults
Brief Title: Can Physical Activities Reduce Postoperative Pain in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 104042
Record Dates: First submitted 2020-01-30; First posted 2020-03-03 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain; Physical Activity
Keywords: postoperative pain; Physical Activity; Non-Physical Activity; Enhanced Recovery After Surgery; Prehabilitation
MeSH Terms: conditions — Pain, Postoperative; Motor Activity

STUDY DESIGN:
Intervention Model Description: latent growth modeling using structural equation model,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity group (Experimental): 1. Investigators employ the recommendations of the American College of Sport Medicine and the World Health Organization for adults to divide our enrolled patients having moderate-intensity as 30-60 min∙d-1 (≥150 min∙wk-1 ) or vigorous-intensity as 20-60 min∙d-1 (≥75 min∙wk-1) for 6-8 weeks preoperatively.
  2. The severity of postoperative pain are measured prospectively at 1, 4, 7, 10 and 24 hours after the surgical operations.
  3. The operations are performed under inhalation general anesthesia with endotracheal intubation or through laryngeal mask.
  Interventions: Procedure: Compare the severity of postoperative pain of the physical activity group Vs non-physical activity group
- non-physical activity group (Experimental): 1. No any moderate-intensity or vigorous-intensity physical activity for our enrolled patients preoperatively.
  2. The severity of postoperative pain are measured prospectively at 1, 4, 7, 10 and 24 hours after the surgical operations.
  3. Various types of operations are performed under inhalation general anesthesia with endotracheal intubation or through laryngeal mask.
  Interventions: Procedure: Compare the severity of postoperative pain of the physical activity group Vs non-physical activity group

INTERVENTIONS:
Procedure: Compare the severity of postoperative pain of the physical activity group Vs non-physical activity group — Compare postoperative pain scores for the physical activity Vs non-physical activity group

SUMMARY:
Recommendation is strong on physical activity (PA) in the prehabilitation of Enhanced Recovery After Surgery (ERAS) for various types of surgeries. The evidence is however weak regarding ERAS protocols. Many studies have showed that physical exercise and PA have hypoalgesic effects on healthy individuals and they have better pain tolerance too. Here the investigators study changes in postoperative pain and postoperative nausea and vomiting for various types of surgical patients after performing preoperative PA at moderate or vigorous intensity Vs non-preoperative PA patients.

DETAILED DESCRIPTION:
The US Institute of Medicine revealed that 80% of patients receiving surgery have reported postoperative pain with 88% of them at moderate, severe, or extreme levels. Opioids for postoperative pain are commonly administered to relieve moderate to severe pain, therefore, the postoperative nausea and vomiting (PONV) incidence will be increased.

ERAS is a prevalent policy that combines evidence-based perioperative care to accelerate surgical recovery, Anesthesiologists are involved in many perioperative ERAS elements of patients in terms of evaluation and implementation: e.g., like prehabilitation via education of physical and core muscles training on the pain management clinic, perioperative multi-modal pain management and multi-modal anti-emetic prophylaxis against PONV.

The overarching aim of multimodal structured prehabilitation programs is to increase, for instance, the cardiopulmonary and musculoskeletal preoperative functional reserve, leading to better postoperative functional recovery and a reduced incidence of complications.

Better ischemic pain tolerance is well documented after combined moderate-and vigorous-intensity aerobic exercise for healthy individuals and acute exercise also has hypoalgesic effects.Unfortunately, these physical activity (PA) researchers have not evaluated specifically effects on postoperative pain and PONV.

The goal of our study is to determine the relationship between preoperative PA on postoperative pain and PONV for different types of surgery.

METHODS:

This is a single center, randomized prospective (preoperative PA patients group vs preoperative non-PA patients group) trial. Information on the incidence and severity of pain and PONV of each patient are periodically recorded at time-points of 1, 4, 7, 10 and 24 hours after various types of surgical operation. Our study was aimed to determine beneficial effects on postoperative pain and PONV for patients after performing preoperative PA for 6 to 8 weeks vs non-PA patients. The investigators employed the recommendations of the American College of Sport Medicine and the World Health Organization for adults to divide our PA patients group into moderate-intensity as 30-60 min∙d-1 (≥150 min∙wk-1 ) and vigorous-intensity as 20-60 min∙d-1 (≥75 min∙wk-1). The severity of postoperative pain and PONV were measured at 1, 4, 7, 10 and 24 hours after the surgical operations for the PA patients group and the non-PA patients group by one of the three registered nurses of our Anesthesiology Department. The severity of postoperative pain were recorded by using 0-10 Numeric Rating Scale and postoperative nausea and vomiting after surgeries were measured by using 5 points Likert Scale (1-5) to record the severity of postoperative pain and PONV after different types of surgery.

The operations were performed under general anesthesia (GA) with endotracheal intubation or inhalation through laryngeal mask.

The procedures of GA will be discussed and decided by one of our anesthesiologists of the Chia-Yi Christian Hospital together with patients/caregivers at the Pre-Anesthesia Consultation Clinic. We used the American Society of Anesthesiologists physical status scoring system for risk stratification, the approaches of Apfel's preventive strategy of postoperative nausea and vomiting prophylaxis, perioperative multi-modal pain management in addition to other appropriate elements in ERAS. PONV defined as nausea, vomiting or retching within 24 h of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥18 y/o
2. Enrolled in-patients
3. Patients are scheduled to undergo various operations.
4. The surgeries are expected to last ≥60 minutes
5. Endotracheal intubation or laryngeal mask inhalation general anesthesia.

Exclusion Criteria:

1. Patients will transferred to the intensive care unit after operations.
2. American Society of Anesthesiology physical status ≥4
3. poorly controlled diabetic mellitus (HA1c ≥9)
4. prolonged corrected QT interval (male ≥0.45 sec, female ≥0.47 sec)
5. Allergy to any opioids (i.e., morphine, fentanyl, pethidine and others) and nonopioids (i.e., selective or nonselective NSAIDs and acetaminophen)
6. Allergy to dexamethasone, granisetron, droperidol, metoclopramide used for prevention of postoperative nausea and vomiting
7. Deaf or unable to speak/understand Taiwanese or Mandarin
8. Failed to recall or uncertain on how many days/times they had spent doing moderate or vigorous physical activity on recent 6 to 8 weeks before receiving surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
The beneficial effect of physical activity on postoperative pain after various types of surgeries | 2 years and 6 months
  1. The pain scores different of the physical activity (PA) Vs non-physical activity (non-PA) groups are using the numeric pain rating scale (NRS) with 1 represent no pain and 5 represent the worst possible pain.
  2. The severity of postoperative pain will be measured prospectively by using NRS at different postoperative time points (i.e. 1, 4, 7, 10, and 24 hour) for comparing the postoperative pain different between PA and non-PA patients.

CONTACTS AND LOCATIONS:
Overall Officials: Wui-Chiu Mui, M.D., MBA, Principal Investigator — Chiayi Christian Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pogatzki-Zahn EM, Segelcke D, Schug SA. Postoperative pain-from mechanisms to treatment. Pain Rep. 2017 Mar 15;2(2):e588. doi: 10.1097/PR9.0000000000000588. eCollection 2017 Mar. PMID 29392204
- [Background] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Milliken D, Schofield N. Understanding Prehabilitation. Anaesthesia 2018; Tutorial Of The Week 394: 1-5.
- [Background] Jones MD, Booth J, Taylor JL, Barry BK. Aerobic training increases pain tolerance in healthy individuals. Med Sci Sports Exerc. 2014 Aug;46(8):1640-7. doi: 10.1249/MSS.0000000000000273. PMID 24504426
- [Background] Naugle KM, Riley JL 3rd. Self-reported physical activity predicts pain inhibitory and facilitatory function. Med Sci Sports Exerc. 2014 Mar;46(3):622-9. doi: 10.1249/MSS.0b013e3182a69cf1. PMID 23899890
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Hu L, Bentler PM. Cutoff criteria for fit indexes in covariance structure analysis: conventional criteria versus new alternatives. Structural Equation Modeling 1999; 6(1): 1-55